CLINICAL TRIAL: NCT03681015
Title: A Multicenter, Prospective, Longitudinal, Digital Assessment Study of Disease Progression in Subjects with Early, Untreated Parkinson Disease
Brief Title: Wearable Assessments in the Clinic and Home in PD
Acronym: WATCH-PD
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: Biogen (Industry); Takeda (Industry)
Responsible Party: Principal Investigator, Ray Dorsey, Professor, University of Rochester
Other Study IDs: WPD-01
Record Dates: First submitted 2018-09-10; First posted 2018-09-21 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2022-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort 1 - Parkinson's Disease Participants: Volunteers will be women and men with early, untreated Parkinson disease.
- Cohort 2 - Control Participants: Participants will be women and men without PD.

SUMMARY:
The purpose of this study is to evaluate disease progression in persons with early Parkinson disease, as assessed by digital and electronic sensor data collection to be correlated with typical clinical assessments.

DETAILED DESCRIPTION:
Subjects will be evaluated via both in-clinic and at-home assessments. The in-clinic assessments are designed to compare the ability of current Parkinson disease clinical trial measures with the ability of mobile and wearable devices to detect disease progression in the early stage of disease. The at-home assessments are designed to determine the feasibility of motor and non-motor assessments of disease progression using a commercially available wearable device/mobile application platform and to determine how this data compares with traditional clinical measures.

ELIGIBILITY:
Cohort 1 (PD Participants) Inclusion Criteria:

1. Able to give written informed consent, as determined by the investigator.
2. Subjects must have at least two of the following: resting tremor, bradykinesia, rigidity (must have either resting tremor or bradykinesia as one of two symptoms); OR either asymmetric resting tremor or asymmetric bradykinesia.
3. Screening dopamine transporter (DAT) SPECT scan is consistent with dopamine transporter deficit.
4. A diagnosis of Parkinson disease for 2 years or less at screening.
5. Modified Hoehn and Yahr stage <=II at screening.
6. Not expected to require PD medication for at least 6 months from baseline (includes dopaminergics, MAO-B inhibitors, and anti-cholinergics used to treat PD-related symptoms).
7. Male or female age 30 years or older at time of PD diagnosis.
8. Female subjects of childbearing potential must agree to be using highly effective contraception within 30 days prior to DaTscan (e.g., oral contraceptives, a barrier method of birth control (e.g., condoms with contraceptive foam, diaphragm with contraceptive jelly), intrauterine device, partner with vasectomy or sexual abstinence).
9. Male subjects who are fertile and have a partner of childbearing potential must agree to use reliable contraception for 14 days following the administration of DaTscanTM (e.g., condoms with contraceptive foam or sexual abstinence).
10. Fluent in English and able to read.
11. Able to perform all study activities (including walking tasks and timed up and go)
12. Willingness and ability to comply with study requirements.

Cohort 1 (PD Participants) Exclusion Criteria

1. A diagnosis of atypical parkinsonism, drug-induced parkinsonism, essential tremor, primary dystonia or other diagnoses that explain symptoms other than PD.
2. History of PD-related freezing episodes or falls.
3. A diagnosis of a significant CNS disease other than PD; history of repeated head injury; history of epilepsy or seizure disorder other than febrile seizures as a child that would interfere with ability to perform study assessments.
4. History of a brain magnetic resonance imaging (MRI) scan indicative of clinically significant abnormality as determined by the investigator.
5. Concomitant disease, condition, medication, or laboratory abnormality that, in the opinion of the investigator, could interfere with study conduct or analysis, or pose an unacceptable risk to the participant. This could include neurologic, orthopedic or cardiovascular diseases.
6. Has taken levodopa, dopamine agonists, MAO B inhibitors, amantadine, anticholinergics or other medication for the treatment of PD or tremor within 60 days prior to baseline, or for more than a total of 60 days.
7. Is taking medication for the treatment of tremor at the baseline visit. If taking medication for tremor at the screening visit, this medication must be stopped at least 14 days prior to baseline. If taking a tremor medication for another indication (e.g.

   hypertension, neuropathy), the medication can be continued during the study.
8. For subjects taking any drugs that might interfere with dopamine transporter SPECT imaging (modafinil, bupropion, methylphenidate, neuroleptics, metoclopramide, alpha methyldopa, reserpine, or amphetamine derivative) must be willing and able from a medical standpoint to withhold the medication for at least 14 days prior to screening DaTscan imaging.
9. Montreal Cognitive Assessment (MoCA) score < 24 at screening.
10. Is pregnant (or is planning to become pregnant during the study period) or lactating (includes a negative urine (or serum if required by site) pregnancy test on day of screening scan prior to injection of DaTscanTM
11. Known hypersensitivity to DaTscanTM or any of its excipients
12. Body habitus that would impede completion of DaTscanTM (subject weight above 158 kg should be discussed with the Clinical Monitor)
13. Resides in a nursing home or assisted care facility.
14. Use of investigational drugs (other than imaging agents) or devices (other than mobile/wearable devices used in this study) within 60 days or 5 half-lives of study agent prior to baseline and during the study period.

Cohort 2 (Control Participants) Inclusion Criteria:

1. Able to give written informed consent, as determined by the investigator.
2. Male or female age 30 years or older at time of PD diagnosis.
3. Fluent in English and able to read.
4. Able to perform all study activities (including walking tasks and timed up and go)
5. Willingness and ability to comply with study requirements.

Cohort 2 (Control Participants) Exclusion Criteria:

1. A diagnosis of atypical parkinsonism, drug-induced parkinsonism, essential tremor, primary dystonia or other diagnoses that explain symptoms other than PD.
2. History of PD-related freezing episodes or falls.
3. A diagnosis of a significant CNS disease other than PD; history of repeated head injury; history of epilepsy or seizure disorder other than febrile seizures as a child that would interfere with ability to perform study assessments.
4. History of a brain magnetic resonance imaging (MRI) scan indicative of clinically significant abnormality as determined by the investigator.
5. Concomitant disease, condition, medication, or laboratory abnormality that, in the opinion of the investigator, could interfere with study conduct or analysis, or pose an unacceptable risk to the participant. This could include neurologic, orthopedic or cardiovascular diseases.
6. Has taken levodopa, dopamine agonists, MAO B inhibitors, amantadine, anticholinergics or other medication for the treatment of PD or tremor within 60 days prior to baseline, or for more than a total of 60 days.
7. Is taking medication for the treatment of tremor at the baseline visit. If taking medication for tremor at the screening visit, this medication must be stopped at least 14 days prior to baseline. If taking a tremor medication for another indication (e.g. hypertension, neuropathy), the medication can be continued during the study.
8. Montreal Cognitive Assessment (MoCA) score < 24 at screening.
9. Resides in a nursing home or assisted care facility.
10. Use of investigational drugs (other than imaging agents) or devices (other than mobile/wearable devices used in this study) within 60 days or 5 half-lives of study agent prior to baseline and during the study period.
11. Is pregnant (or is planning to become pregnant during the study period) or lactating.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohort 1 (PD Participants): Male and female subjects with early, untreated Parkinson's disease, aged 30 years or older at time of disease diagnosis
  Cohort 2 (Control Participants): Male and female subjects without Parkinson's disease, aged 30 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2022-02-21 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Change and variability in inertial sensor-derived measures of motor function from baseline to 12 months during performance of the MDS-UPDRS part 3 motor exam. | 12 months
  Features will be extracted from continuous accelerometer and gyroscope signals, obtained via a set of body-worn inertial sensors, during performance of the MDS-UPDRS part 3, and the change and variability of these features will be assessed.
Correlations between inertial sensor-derived measures of motor function and clinician ratings during performance of the MDS-UPDRS part 3 and total exam at baseline, 1, 3, 6, 9, and 12 months. | 12 months
  Features extracted from continuous accelerometer and gyroscope signals recorded during each relevant component of the UPDRS part 3 will be correlated with corresponding clinician ratings to quantify the relationship between these measures.

SECONDARY OUTCOMES:
Correlations between sensor-derived measures of motor function (accelerometer, gyroscope) and patient-reported outcomes measured by MDS-UPDRS parts 1b and 2 at baseline, 1, 3, 6, 9, and 12 months. | 12 months
  Features extracted from continuous accelerometer and gyroscope signals, recorded during the UPDRS part 3 will be correlated with scores on the UPDRS 1b and 2 subtests to examine how sensor-derived measures relate to patient reported activities of daily living and quality of life.
Correlations between sensor-derived measures of motor function (accelerometer, gyroscope) and patient-reported outcomes measured by PDQ-8 at baseline, 1, 3, 6, 9, and 12 months. | 12 months
  Features extracted from continuous accelerometer and gyroscope signals, recorded during the UPDRS part 3 will be correlated with scores on the PDQ-8 to examine how sensor-derived measures relate to patient reported quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Earl R Dorsey, MD MBA, Principal Investigator — University of Rochester
Locations (17):
- United States (17):
  - Banner Sun Research Institute, Sun City, Arizona
  - University of California San Francisco, San Francisco, California
  - University of Colorado Denver, Aurora, Colorado
  - University of South Florida, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Cleveland Clinic Nevada, Las Vegas, Nevada
  - Northwell Health, Great Neck, New York
  - NYU Langone Health, New York, New York
  - University of Rochester, Rochester, New York
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Sentara Clinical Research, Virginia Beach, Virginia